CLINICAL TRIAL: NCT01392885
Title: Brain Health: Effects of Exercise on Hippocampal Volume and Memory Deficits in Persons With Schizophrenia
Brief Title: Brain Health and Exercise in Schizophrenia
Acronym: PEHP
Status: Recruiting | Type: Observational
Sponsor: BC Mental Health and Addictions Research Institute (Other Government)
Collaborators: University of British Columbia (Other); Simon Fraser University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Donna Lang, PhD, Dr. Donna J. Lang, PhD, BC Mental Health and Addictions Research Institute
Other Study IDs: 231233-BSB
Record Dates: First submitted 2011-06-21; First posted 2011-07-13 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Poor Memory
Keywords: Schizophrenia; Schizoaffective Disorder; Brain Health; Exercise; Mental Health; Poor memory
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Memory Disorders; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — No Biospecimens to be retained
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the effects of aerobic exercise on hippocampal volumes and severity of psychotic symptoms in a population of psychosis patients compared to healthy age/gender matched volunteers. Psychosis patients often suffer from a number of cognitive difficulties, including poor memory function, poor problem-solving capacity and difficulties with attention and concentration. Poor fitness and associated neurovascular deficits may arise from various sources, including poor mental health, adverse side effects of antipsychotic medications and independent cardiovascular deficits that may be due to neurodevelopmental abnormalities in patients with schizophrenia. These factors are likely contributing to markedly increased stroke risk and early mortality. These problems are not well addressed by current clinical treatments, nor is neurovascular stroke risk readily or accurately detected in clinic.In contrast, evidence from aging research strongly suggests that increased cardiovascular fitness may provide numerous cognitive benefits by promoting brain growth, particularly in the frontal lobes and the hippocampi, while reducing the risk of stroke. The current study will measure the effects of aerobic exercise on brain volumes in a population of chronic psychosis patients to determine if 1) hippocampal volumes increase in response to exercise and 2) if parallel improvements in cognitive functioning occur. Additionally, baseline and follow-up stroke risk will be assessed using a novel non-invasive approach of retinal imaging to determine the presence of underlying neurovascular pathology.

DETAILED DESCRIPTION:
This is a 12-week, randomized trial with two parallel groups. Throughout the trial, subjects will be treated on their prescribed dose of medication. Once informed consent is obtained, subjects and healthy volunteers will be randomly assigned to either an aerobic or a resistance exercise program (N = 30 per diagnostic group in each of two exercise conditions). Patients will continue to receive their antipsychotics and other prescribed medications. Healthy volunteer data will be used to establish normal exercise-induced neuroplasticity in a non-psychiatric, non-medicated population and to establish differences in retinal vessel integrity between patients and healthy volunteers. All training will be conducted at the UBC Hospital and at dedicated exercise training facilities at the University of British Columbia. All fitness assessments (based on the initial 6-minute walk test) and exercise sessions will be monitored by trained research assistants (RAs) under the guidance of the Canadian Society for Exercise Physiology-Certified Exercise Physiologists (CSEP-CEPs). The RAs will receive pre-study exercise training from the CSEP-CEPs. During the course of the study, the training intensity will be changed according to the individual participant's response and needs via the CSEP-CEPs and RAs.

Clinical data (current medications, current diagnoses, symptom profiles, resting heart rate, blood pressure, weight) will be collected on the hospital wards at baseline and follow-up. Neuroimaging and retinal imaging will be ascertained at the UBC MRI Research Centre at baseline and follow-up. Concurrent baseline assessments of executive functioning, memory capacity and crystallized IQ will be performed at baseline. Cognitive measures, excluding IQ, will be re-assessed at follow-up. Follow-up measures will only be collected in cases were patients are still available and willing to participate in study activities.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years
* Able to provide written, informed consent in English
* Patients may be on prescribed medications
* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Normal visual acuity (or normal visual acuity achievable with corrective lenses)
* Physical ability to be engaged in a regular exercise program

Exclusion Criteria:

* A history of organic disorders (dementia, severe head injury, or developmental disorders such as autism, mental retardation, Down's Syndrome)
* A current DSM-IV diagnosis of substance dependence (during prior 12 months, excluding tobacco)
* Any history of DSM-IV diagnoses (Axis I) for other psychiatric disorders
* History of angina, heart attack or transient ischemic attacks
* Non-independent mobility or limb prostheses
* A history of severe head injury leading to loss of consciousness for > 5 minutes
* Contra-indications for neuroimaging (metal implants, non-removable orthodontic devices, severe claustrophobia, pregnancy, or surgeries within the previous 6 months)
* Currently already enrolled in a regular exercise program

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sixty in-patients with chronic schizophrenia will be recruited at UBC Hospital and 60 age and gender-matched healthy (asymptomatic) community volunteers will be recruited through local community paper advertisements or posters at local community centres.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Increase hippocampal volume with aerobic training in schizophrenic and healthy volunteers. | Base-line, 8 and 12 weeks
  Hippocampal volumes will be measured from structural MRI scans. T1-weighted 3D SPGR (spoiled gradient recalled) and high-resilution T2- weighted structural images will be obtained for the purposes of volumetric assessment of the hippocampi and the whole brain

SECONDARY OUTCOMES:
Increases in hippocampal volumes will be positively associated with improvements in working memory performance in schizophrenia. | Baseline, Week 4, 8 and 12.
  The Hopkins Verbal Learning Test (HVLT), will be used to assess memory function. Multiple versions of the HVLT exist (12) so practice effects will be minimized. The Rey-Osterrieth Complex Figure Test (ROCF), in which subjects are asked to reproduce a complex line drawing from memory, will be used to assess attention and working memory.

CONTACTS AND LOCATIONS:
Overall Officials: Donna J Lang, PhD, Principal Investigator — University of British Columbia, Dept. of Radiology; William G Honer, Professor, Study Chair — University of British Columbia, Dept of Psychiatry; Allen Thornton, Unspecified, Study Chair — Simon Fraser University; Darren Warburton, Ass. Prof, Study Chair — University of British Columbia, Dept. of Human Kinetics; Alexandra T Vertinsky, Clin. Instr., Study Chair — University of British Columbia, Dept. of Radiology; Alexander Rauscher, Ass. Prof., Study Chair — University of British Columbia, Dept. of Radiology
Locations (1):
- UBC Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Woodward ML, Gicas KM, Warburton DE, White RF, Rauscher A, Leonova O, Su W, Smith GN, Thornton AE, Vertinsky AT, Phillips AA, Goghari VM, Honer WG, Lang DJ. Hippocampal volume and vasculature before and after exercise in treatment-resistant schizophrenia. Schizophr Res. 2018 Dec;202:158-165. doi: 10.1016/j.schres.2018.06.054. Epub 2018 Jun 29. PMID 30539767
- [Derived] Kim DD, Lang DJ, Warburton DER, Woodward ML, White RF, Barr AM, Honer WG, Procyshyn RM. Heart-rate response to alpha2-adrenergic receptor antagonism by antipsychotics. Clin Auton Res. 2017 Dec;27(6):407-410. doi: 10.1007/s10286-017-0444-4. Epub 2017 Jul 3. PMID 28674870